CLINICAL TRIAL: NCT03355209
Title: A Two-Part Study of ZX008 in Children and Adults With Lennox-Gastaut Syndrome (LGS); Part 1: A Randomized, Double-blind, Placebo-controlled Trial of Two Fixed Doses of ZX008 (Fenfluramine Hydrochloride) Oral Solution as Adjunctive Therapy for Seizures in Children and Adults With LGS, Followed by Part 2: An Open-label Extension to Assess Long-Term Safety of ZX008 in Children and Adults With LGS
Brief Title: A Study to Investigate the Efficacy and Safety of ZX008 (Fenfluramine Hydrochloride) as an Adjunctive Therapy in Children and Adults With Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX008-1601; 2017-002628-26 (EudraCT Number)
Record Dates: First submitted 2017-06-19; First posted 2017-11-28 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Lennox Gastaut Syndrome
Keywords: LGS
MeSH Terms: conditions — Lennox Gastaut Syndrome

STUDY DESIGN:
Intervention Model Description: Part 1: Double-Blind ZX008 - (0.2 mg/kg/day or 0.8mg/kg/day) or Placebo and Part 2: Open-Label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1: Double-Blind Part 2: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ZX008 0.2 or 0.8 mg/kg/day (Experimental): Part 1: ZX008 is supplied as an oral solution. Subjects will be randomized to receive 1 of 2 doses of ZX008 0.2 mg/kg/day or 0.8 mg/kg/day.
  Interventions: Drug: ZX008 0.2 or 0.8 mg/kg/day
- Matching Placebo (Placebo Comparator): Part 1: Matching ZX008 placebo is supplied as an oral solution.
  Interventions: Drug: Matching Placebo
- Open-Label (Experimental): Part 2: ZX008 is supplied as an oral solution. Study medication will be administered twice a day (BID) in equally divided doses.
  Interventions: Drug: ZX008 0.2 or 0.8 mg/kg/day

INTERVENTIONS:
Drug: ZX008 0.2 or 0.8 mg/kg/day — ZX008 drug product is an oral aqueous solution of fenfluramine hydrochloride. The product is sugar free and is intended to be compatible with a Ketogenic Diet.
  Arms: Open-Label; ZX008 0.2 or 0.8 mg/kg/day
Drug: Matching Placebo — Placebo will be administered twice a day (BID) in equally divided doses.
  Other Names: Placebo Comparator
  Arms: Matching Placebo

SUMMARY:
This is a two-part, multicenter, double-blind, parallel-group, placebo controlled study to evaluate the effect of ZX008 when used as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with Lennox-Gastaut syndrome (LGS).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or non-pregnant, non-lactating female, age 2 to 35 years, inclusive as of the day of the Screening Visit.
* Clinical diagnosis of Lennox-Gastaut syndrome, where seizures that result in drops are not completely controlled by current antiepileptic treatments.
* Onset of seizures at 11 years of age or younger.
* Abnormal cognitive development.
* Must be receiving at least 1 concomitant AED and up to 4 concomitant anti-epileptic treatments.

Key Exclusion Criteria:

* Etiology of seizures is a degenerative neurological disease.
* History of hemiclonic seizures in the first year of life.
* Subject only has drop seizures in clusters, where individual seizures cannot be counted reliably.
* Pulmonary arterial hypertension.
* Current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke.
* Receiving concomitant therapy with: centrally-acting anorectic agents; monoamineoxidase inhibitors; any centrally-acting compound with clinically appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; atomoxetine, or other centrally-acting noradrenergic agonist; cyproheptadine.
* Taking felbamate for less than 1 year prior to screening and/or does not have stable liver function and hematology laboratory tests, and/or the dose has not been stable for at least 60 days prior to the Screening Visit.
* Currently receiving an investigational product.
* Institutionalized in a general nursing home (ie, in a facility that does not specialize in epilepsy care).
* A clinically significant condition, or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to the Screening Visit, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 296 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (72):
- United States (30):
  - Ep0214 107, Tucson, Arizona
  - Ep0214 144, Los Angeles, California
  - Ep0214 101, San Francisco, California
  - Ep0214 103, Aurora, Colorado
  - Ep0214 149, Washington D.C., District of Columbia
  - Ep0214 115, Gulf Breeze, Florida
  - Ep0214 104, Miami, Florida
  - Ep0214 141, Orlando, Florida
  - Ep0214 121, Orlando, Florida
  - Ep0214 117, Atlanta, Georgia
  - Ep0214 110, Chicago, Illinois
  - Ep0214 140, Bethesda, Maryland
  - Ep0214 112, Boston, Massachusetts
  - Ep0214 136, Grand Rapids, Michigan
  - Ep0214 147, Royal Oak, Michigan
  - Ep0214 109, Rochester, Minnesota
  - Ep0214 132, Saint Paul, Minnesota
  - Ep0214 105, Hackensack, New Jersey
  - Ep0214 118, Livingston, New Jersey
  - Ep0214 150, Hartsdale, New York
  - Ep0214 142, New York, New York
  - Ep0214 131, Cleveland, Ohio
  - Ep0214 143, Portland, Oregon
  - Ep0214 120, Philadelphia, Pennsylvania
  - Ep0214 139, York, Pennsylvania
  - Ep0214 146, Dallas, Texas
  - Ep0214 126, Fort Worth, Texas
  - Ep0214 145, San Antonio, Texas
  - Ep0214 106, Salt Lake City, Utah
  - Ep0214 125, Tacoma, Washington
- Australia (2):
  - Ep0214 301, Heidelberg
  - Ep0214 302, South Brisbane
- Belgium (3):
  - Ep0214 802, Brussels
  - Ep0214 803, Brussels
  - Ep0214 801, Edegem
- Canada (2):
  - Ep0214 204, Toronto
  - Ep0214 201, Vancouver
- Ep0214 701, Dianalund, Denmark
- France (6):
  - Ep0214 1004, Bordeaux
  - Ep0214 1006, Bron
  - Ep0214 1005, Lille
  - Ep0214 1007, Marseille
  - Ep0214 1001, Paris
  - Ep0214 1002, Paris
- Germany (6):
  - Ep0214 902, Bielefeld
  - Ep0214 906, Freiburg im Breisgau
  - Ep0214 905, Jena
  - Ep0214 908, Kiel
  - Ep0214 903, Radeberg
  - Ep0214 901, Vogtareuth
- Italy (5):
  - Ep0214 1211, Bologna
  - Ep0214 1201, Florence
  - Ep0214 1204, Genova
  - Ep0214 1206, Roma
  - Ep0214 1208, Roma
- Japan (8):
  - Ep0214 1510, Fukuoka
  - Ep0214 1505, Niigata
  - Ep0214 1501, Okayama
  - Ep0214 1507, Osaka
  - Ep0214 1504, Ōmura
  - Ep0214 1508, Sapporo
  - Ep0214 1506, Shinjuku-ku
  - Ep0214 1502, Shizuoka
- Ep0214 1604, Guadalajara, Mexico
- Ep0214 1401, Zwolle, Netherlands
- Poland (2):
  - Ep0214 1702, Bydgoszcz
  - Ep0214 1701, Krakow
- Spain (4):
  - Ep0214 1105, Barcelona
  - Ep0214 1107, Barcelona
  - Ep0214 1101, Mirasierra
  - Ep0214 1102, Pamplona
- Ep0214 502, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Derived] Knupp KG, Scheffer IE, Ceulemans B, Sullivan JE, Nickels KC, Lagae L, Guerrini R, Zuberi SM, Nabbout R, Riney K, Shore S, Agarwal A, Lock M, Farfel GM, Galer BS, Gammaitoni AR, Davis R, Gil-Nagel A. Efficacy and Safety of Fenfluramine for the Treatment of Seizures Associated With Lennox-Gastaut Syndrome: A Randomized Clinical Trial. JAMA Neurol. 2022 Jun 1;79(6):554-564. doi: 10.1001/jamaneurol.2022.0829. PMID 35499850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in November 2017 and concluded in May 2024. Cohort A included participants enrolled at sites in North America, Europe, and Australia. Cohort B included participants enrolled at sites in Japan only.
Pre-assignment Details: The Participant Flow refers to the All Enrolled Participants Set for Part 1 and OLE Safety Population for Part 2 of the study. As planned, Part 2 summaries were presented by the participant's Part 1 treatment groups (placebo, ZX008 0.2 mg/kg/day, ZX008 0.8 mg/kg/day).
Groups:
- Cohort A: Placebo: Part 1: Participants received matching placebo as an oral solution, twice a day (bid) over 2 weeks of Titration Period and an additional 12 weeks of Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days. In Part 2 (OLE Period): Participants initially received ZX008 0.2 mg/kg/day for 1 month. After 1 month, the Investigator could adjust the dose if needed. Participants received ZX008 for up to 12 months in OLE Period.
- Cohort A: ZX008 0.2 mg/kg/Day: Part 1: Participants received ZX008 0.2 milligram per kilogram per day (mg/kg/day) during the 2-week Titration. Following titration, participants received ZX008 0.2 mg/kg/day as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days. In Part 2 (OLE Period): Participants initially received ZX008 0.2 mg/kg/day for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Participants received ZX008 for up to 12 months in OLE Period.
- Cohort A: ZX008 0.8 mg/kg/Day: Part 1: Participants were titrated to their blinded randomized dose of ZX008 over the 2-week Titration from 0.2 mg/kg/day to ZX008 0.8 mg/kg/day (or a maximum dose of 30 mg/day or 20 mg/day for participants taking concomitant stiripentol [STP]). Following titration, participants continued to receive the randomized dose of ZX008 as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days. In Part 2 (OLE Period): Participants initially received ZX008 0.2 mg/kg/day for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Participants received ZX008 for up to 12 months in OLE Period.
- Cohort B: Placebo: Part 1: Participants received matching placebo as an oral solution, bid over 2 weeks of Titration Period and an additional 12 weeks of Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days. In Part 2 (OLE Period): Participants initially received ZX008 0.2 mg/kg/day for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Participants received ZX008 for up to 12 months in OLE Period. Participants who completed 12 months OLE Period had option to receive ZX008 for up to 72 months, or until ZX008 is approved in the participant's country.
- Cohort B: ZX008 0.2 mg/kg/Day: Part 1: Participants received ZX008 0.2 mg/kg/day during the 2-week Titration. Following titration, participants received ZX008 0.2 mg/kg/day as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days. In Part 2 (OLE Period): Participants initially received ZX008 0.2 mg/kg/day for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Participants received ZX008 for up to 12 months in OLE Period. Participants who completed 12 months OLE Period had option to receive ZX008 for up to 72 months, or until ZX008 is approved in the participant's country.
- Cohort B: ZX008 0.8 mg/kg/Day: Part 1: Participants were titrated to their blinded randomized dose of ZX008 over the 2-week Titration from 0.2 mg/kg/day to ZX008 0.8 mg/kg/day (or a maximum dose of 30 mg/day or 20 mg/day for participants taking concomitant STP). Following titration, participants continued to receive the randomized dose of ZX008 as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days. In Part 2 (OLE Period): Participants initially received ZX008 0.2 mg/kg/day for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Participants received ZX008 for up to 12 months in OLE Period. Participants who completed 12 months OLE Period had option to receive ZX008 for up to 72 months, or until ZX008 is approved in the participant's country.
Period: Part 1: Double-Blind Period
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Started | 87 | 89 | 87 | 11 | 11 | 11
Completed (Participants who completed visits up to Week 14 or transitioned early to Part 2) | 86 | 83 | 81 | 11 | 10 | 11
Not Completed | 1 | 6 | 6 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 4 | 4 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0 | 0
Period: Part 2:Open-Label Extension (OLE) Period
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Started | 86 | 83 | 78 | 11 | 10 | 11
Completed | 61 | 51 | 46 | 5 | 1 | 5
Not Completed | 25 | 32 | 32 | 6 | 9 | 6
Not completed — Adverse Event | 5 | 5 | 3 | 0 | 1 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 13 | 21 | 23 | 0 | 0 | 1
Not completed — Switching to commercial ZX008 | 0 | 0 | 0 | 5 | 6 | 3
Not completed — Withdrawal by Subject | 6 | 5 | 4 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Rollover into ZX008-1900 | 1 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to Safety Population which consisted of all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day | Total
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (7.71) | 13.4 (7.79) | 13.4 (7.28) | 18.5 (7.78) | 20.1 (7.79) | 18.5 (7.94) | 14.3 (7.76)
Age, Customized [Count of Participants; unit: Participants]
  2 - < 12 years | 32 | 41 | 37 | 2 | 3 | 2 | 117
  12 - < 18 years | 29 | 23 | 25 | 5 | 2 | 3 | 87
  18 - 35 years | 26 | 25 | 25 | 4 | 6 | 6 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 33 | 5 | 2 | 2 | 126
  Male | 46 | 46 | 54 | 6 | 9 | 9 | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 71 | 67 | 70 | 0 | 0 | 0 | 208
  Black or African American | 4 | 5 | 3 | 0 | 0 | 0 | 12
  Asian | 2 | 3 | 4 | 11 | 11 | 11 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Reported | 6 | 11 | 7 | 0 | 0 | 0 | 24
  Unknown | 2 | 2 | 2 | 0 | 0 | 0 | 6
  Multiple | 2 | 0 | 1 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 14 | 0 | 0 | 0 | 51
  Not Hispanic or Latino | 65 | 58 | 66 | 11 | 11 | 11 | 222
  Not Reported | 6 | 10 | 7 | 0 | 0 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percent Change From Baseline in the Frequency of Seizures That Result in Drops (ESC-confirmed) in the Combined Titration and Maintenance Period (T+M) in the ZX008 0.8 mg/kg/Day Group Compared to the Placebo Group
Description: Percent change in frequency of seizures that result in drops (DSF: drop seizure frequency) per 28 days between the combined Titration and Maintenance (T+M) and Baseline. The percent change from Baseline DSF was calculated as the change in DSF between T+M and Baseline / DSF during Baseline* 100. The seizure types included in the count were: atonic, tonic, tonic/atonic, generalized tonic-clonic, and secondarily generalized tonic-clonic seizures resulting in drops.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: The Modified Intent-to-Treat (mITT) Population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 87 | 11 | 11
percent change | -7.59 [-100.0 to 557.1] | -26.49 [-95.2 to 402.1] | -17.89 [-97.3 to 61.8] | -34.52 [-69.4 to 45.5]
Statistical Analysis 1: Comparison: Cohort A: Placebo vs Cohort A: ZX008 0.8 mg/kg/Day; Test type: Superiority; p = 0.0008, Wilcoxon (Mann-Whitney); Median Difference (A-P) = -19.88, 95% CI 2-sided [-31.02 to -8.74] — Hodges-Lehmann (HL) method

2. Primary Outcome: Part 2: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) was defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of investigational product, or whether considered related to the investigational product. A TEAE in Part 2 was defined as any AE with an onset on or after the first dose in Part 2. AEs with onset in Part 1 that are ongoing in Part 2 were not included in the count of AEs in Part 2.
Time Frame: From Part 2 Baseline until end of the OLE Period (up to 72 months)
Population: The OLE Safety Population included all participants who received at least 1 dose of ZX008 during the OLE. As pre-specified in study design, participants in Part 2 received individualized optimized treatment (0.2 mg/kg/day to 0.8 mg/kg/day) based on Investigator discretion. Hence overall data for Part 2 is reported.
Measure: Number; unit: percentage of participants
Groups:
- Part 2: Cohort A- Overall: All Cohort A participants who continued in Part 2 received ZX008 0.2 mg/kg/day as an oral solution, twice a day (bid), for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Dose changes were made in maximum increments of 0.2 mg/kg/day, to a maximum of 0.8 mg/kg/day (or 0.5 mg/kg/day for participants taking concomitant STP) but not to exceed a total dose of 30 mg/day (or 20 mg/kg/day for participants taking concomitant STP). Participants received ZX008 for up to 12 months in OLE Period.
- Part 2: Cohort B- Overall: All Cohort B participants who continued in Part 2 received ZX008 0.2 mg/kg/day as an oral solution, twice a day (bid), for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Dose changes were made in maximum increments of 0.2 mg/kg/day, to a maximum of 0.8 mg/kg/day (or 0.5 mg/kg/day for participants taking concomitant STP) but not to exceed a total dose of 30 mg/day (or 20 mg/kg/day for participants taking concomitant STP). Participants received ZX008 for up to 12 months in OLE Period. Participants who completed 12 months OLE Period had option to receive ZX008 for up to 72 months, or until ZX008 is approved in the participant's country.
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 247 | 32
percentage of participants | 83.0 | 96.9

3. Primary Outcome: Part 2: Percentage of Participants With Serious TEAEs
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose: Results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is medically significant.
Time Frame: From Part 2 Baseline until end of the OLE Period (up to 72 months)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Part 2: Cohort A- Overall: All Cohort A participants who continued in Part 2 received ZX008 0.2 milligram per kilogram per day (mg/kg/day) as an oral solution, twice a day (bid), for 1 month. After 1 month at a dose of ZX008 0.2 mg/kg/day, the Investigator could adjust the dose if needed. Dose changes were made in maximum increments of 0.2 mg/kg/day, to a maximum of 0.8 mg/kg/day (or 0.5 mg/kg/day for participants taking concomitant STP) but not to exceed a total dose of 30 mg/day (or 20 mg/kg/day for participants taking concomitant STP). Participants received ZX008 for up to 12 months in OLE Period.
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 247 | 32
percentage of participants | 16.6 | 18.8

4. Secondary Outcome: Part 1: Percent Change From Baseline in the Frequency of Seizures That Result in Drops (ESC-confirmed) in T+M in the ZX008 0.2 mg/kg/Day Group Compared to the Placebo Group
Description: as for outcome 1
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 11 | 11
percent change | -7.59 [-100.0 to 557.1] | -14.16 [-100.0 to 3307.3] | -17.89 [-97.3 to 61.8] | -14.12 [-95.6 to 66.4]
Statistical Analysis 1: Comparison: Cohort A: Placebo vs Cohort A: ZX008 0.2 mg/kg/Day; Test type: Superiority; p = 0.1460, Wilcoxon (Mann-Whitney); Median Difference (A-P) = -10.50, 95% CI 2-sided [-24.99 to 3.99] — Hodges-Lehmann (HL) method

5. Secondary Outcome: Part 1: Percentage of Participants Who Achieve a >=50% Reduction From Baseline in the Frequency of Seizures That Result in Drops Comparing the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: The seizure types included in the count were: atonic, tonic, tonic/atonic, generalized tonic-clonic, and secondarily generalized tonic-clonic seizures resulting in drops. Participants who achieved a >=50% reduction from Baseline in the DSF, ie, a decrease in DSF of at least 50 percentage points per 28 days during Titration and Maintenance Period.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percentage of participants | 10.3 | 28.1 | 25.3 | 9.1 | 36.4 | 36.4
Statistical Analysis 1: Comparison: Cohort A: Placebo vs Cohort A: ZX008 0.2 mg/kg/Day; Test type: Superiority; p = 0.0051, Regression, Logistic; Odds Ratio (OR) = 3.30, 95% CI 2-sided [1.43 to 7.59]
Statistical Analysis 2: Comparison: Cohort A: Placebo vs Cohort A: ZX008 0.8 mg/kg/Day; Test type: Superiority; p = 0.0150, Regression, Logistic; Odds Ratio (OR) = 2.87, 95% CI 2-sided [1.23 to 6.70]

6. Secondary Outcome: Part 1: Percentage of Participants Who Achieve Improvement (Minimally, Much or Very Much Improved) in the CGI-I Scale as Assessed by Principal Investigator Comparing ZX008 0.8 and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: Clinical Global Impression - Improvement (CGI-I) scale measures improvement in the participant's condition from Baseline. The severity of a participant's condition was rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), as follows: 1-very much improved,2-much improved, 3-minimally improved, 4- no change, 5-minimally worse, 6-much worse and 7-very much worse.
Time Frame: At Day 99 (Visit 12)
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available. Here, number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 80 | 85 | 80 | 11 | 11 | 11
percentage of participants | 33.8 | 44.7 | 48.8 | 9.1 | 45.5 | 72.7
Statistical Analysis 1: Comparison: Cohort A: Placebo vs Cohort A: ZX008 0.2 mg/kg/Day; Visit 12; Test type: Superiority; p = 0.1565, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.84 to 2.97]
Statistical Analysis 2: Comparison: Cohort A: Placebo vs Cohort A: ZX008 0.8 mg/kg/Day; Visit 12; Test type: Superiority; p = 0.0567, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.86, 95% CI 2-sided [0.98 to 3.52]

7. Secondary Outcome: Part 1: Percent Change From Baseline in Frequency of All Seizures That Typically Result in Drops in T+M, Whether ESC-confirmed as Drop or Not in the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: Seizures that typically result in drops included all: generalized tonic-clonic seizures [GTC], secondarily generalized tonic-clonic [SGTC], tonic seizures [TS], atonic seizures [AS], and tonic/atonic seizures [TA], whether confirmed by the ESC or not. Seizures that result in a drop were defined as seizures involving the entire body, trunk, or head that led to a fall, injury, slumping in a chair, or the participant's head hitting a surface or that could have led to a fall or injury, depending on the patient's position at the time of the seizure.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: as for outcome 4
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percent change | -8.43 [-100.0 to 557.1] | -11.75 [-100.0 to 3307.3] | -26.28 [-95.2 to 402.1] | -17.89 [-97.3 to 61.8] | -14.12 [-95.6 to 66.4] | -34.04 [-69.4 to 45.5]

8. Secondary Outcome: Part 1: Percent Change From Baseline in the Frequency of All Countable Motor Seizures in T+M in the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: Countable motor seizures included: GTC, SGTC, TS, AS, TA, clonic seizures [CS], hemiclonic seizures [HS], and focal seizures [FS] with clearly observable signs.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: as for outcome 4
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percent change | -8.43 [-80.8 to 497.8] | -11.75 [-100.0 to 3307.3] | -26.28 [-91.9 to 402.1] | -17.89 [-97.3 to 61.8] | -14.12 [-95.6 to 174.1] | -34.04 [-69.4 to 45.5]

9. Secondary Outcome: Part 1: Change From Baseline in the Frequency of All Countable Non-motor Seizures in T+M in the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: Countable non-motor seizures included: focal seizures [FS] without clear observable signs, myoclonic seizures [MS], absence/atypical absence, infantile spasms, epileptic spasms, and other seizures. For each participant, the seizure frequency per 28 days was calculated as the number of seizures recorded during the period, divided by the number of days in the period and multiplied by 28.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: as for outcome 4
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
seizure frequency per 28 days | 0.00 [-338.3 to 364.3] | 0.00 [-418.7 to 675.8] | 0.00 [-364.0 to 2952.7] | -7.16 [-30.3 to 13.1] | 0.00 [-32.3 to 104.8] | 0.00 [-61.6 to 209.5]

10. Secondary Outcome: Part 1: Percent Change From Baseline in the Frequency of All Countable Seizures (Motor and Non-motor) in T+M in the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: Countable motor seizures included: GTC, SGTC, TS, AS, TA, CS, HS, and FS with clearly observable signs. Countable non-motor seizures included: FS without clear observable signs, MS, absence/atypical absence, infantile spasms, epileptic spasms, and other seizures.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: as for outcome 4
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percent change | -9.40 [-85.4 to 497.8] | -23.55 [-100.0 to 882.1] | -21.70 [-91.9 to 224.9] | -17.69 [-97.2 to 61.8] | -20.41 [-87.1 to 826.2] | -13.85 [-64.9 to 63.8]

11. Secondary Outcome: Part 1: Percent Change From Baseline in the Frequency of Seizures That Result in Drops (ESC Confirmed) Between Baseline and the Maintenance Period
Description: The frequency of drop seizures during a given interval was derived from the number and type of events recorded in participant electronic diaries. The seizure types included in the count were: atonic, tonic, tonic/atonic, generalized tonic-clonic, and secondarily generalized tonic-clonic seizures resulting in drops.
Time Frame: During Maintenance Period (12 weeks), compared to Baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
percent change | -7.28 [-100.0 to 516.7] | -18.63 [-100.0 to 964.0] | -27.16 [-100.0 to 643.3] | -18.18 [-99.4 to 66.7] | -12.88 [-100.0 to 239.4] | -45.07 [-77.8 to 52.2]

12. Secondary Outcome: Part 1: Percent Change From Baseline in the Frequency of Seizures That Typically Result in Drops in the Maintenance Period in the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: Seizures that typically result in drops included all: GTC, SGTC, TS, AS, and TA, whether confirmed by the ESC or not.
Time Frame: During Maintenance Period (12 weeks), compared to Baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
percent change | -9.37 [-100.0 to 516.7] | -17.30 [-100.0 to 964.0] | -26.30 [-100.0 to 643.3] | -18.18 [-99.4 to 66.7] | -12.88 [-100.0 to 239.4] | -46.88 [-77.8 to 52.2]

13. Secondary Outcome: Part 1: Percent Change From Baseline in the Frequency of All Countable Motor Seizures in the Maintenance Period in the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: Countable motor seizures included: GTC, SGTC,TS, AS, TA, CS, HS, and FS with clearly observable signs.
Time Frame: During Maintenance Period (12 weeks), compared to Baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
percent change | -10.21 [-81.1 to 439.8] | -17.30 [-100.0 to 964.0] | -28.33 [-100.0 to 643.3] | -18.18 [-99.4 to 66.7] | -12.88 [-100.0 to 472.7] | -46.88 [-77.8 to 52.2]

14. Secondary Outcome: Part 1: Change From Baseline in the Frequency of All Countable Non-motor Seizures in the Maintenance Period in the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: as for outcome 9
Time Frame: During Maintenance Period (12 weeks), compared to Baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
seizure frequency per 28 days | -0.04 [-340.6 to 362.3] | -0.13 [-442.3 to 588.1] | 0.00 [-368.3 to 3219.3] | -4.00 [-30.7 to 15.3] | 0.00 [-37.2 to 192.0] | 0.00 [-86.8 to 250.7]

15. Secondary Outcome: Part 1: Percent Change From Baseline in the Frequency of All Countable Seizures (Motor and Non-motor) in the Maintenance Period in ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: as for outcome 10
Time Frame: During Maintenance Period (12 weeks), compared to Baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
percent change | -9.49 [-85.7 to 439.8] | -27.63 [-100.0 to 211.1] | -23.34 [-100.0 to 254.5] | -18.18 [-99.5 to 66.7] | -20.33 [-95.7 to 1626.7] | -17.68 [-72.3 to 80.5]

16. Secondary Outcome: Part 1: Percent Change From Baseline in Frequency of Countable Seizures That do Not Result in Drops (ESC Confirmed)
Description: Non-drop seizures were defined as any countable seizure types that did not meet the criteria of drop seizures, ie, are classified as CS, HC, FS with or without observable signs, MS, absence/atypical absence, infantile spasms, epileptic spasms, or other; or are seizures of the following classifications that were approved for each participant as non-drop seizure types by the ESC: GTC, SGTC, TS, AS, or TA.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: as for outcome 6
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 70 | 73 | 64 | 8 | 7 | 9
percent change | -26.92 [-100.0 to 5070.3] | -31.32 [-100.0 to 571.8] | -22.68 [-100.0 to 481.3] | -23.38 [-96.9 to 657.1] | 0.27 [-32.3 to 2915.4] | -22.99 [-85.7 to 138.8]

17. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a Worsening From Baseline (ie <=0% Reduction), or >0, >=25%, >=50%, >=75%, 100% Reduction, and "Near Seizure Freedom" Between Baseline and T+M, and Baseline and M, in Seizures That Result in Drops
Description: The seizure types included in the count were: atonic, tonic, tonic/atonic, generalized tonic-clonic, and secondarily generalized tonic-clonic seizures resulting in drops. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during T+M); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during combined T+M Period and Maintenance Period were reported.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]; During Maintenance Period (12 weeks), compared to Baseline
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available. Here, Number Analyzed included those participants who were evaluable at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percentage of participants
  Worsening or No Change (T+M) | 37.9 | 34.8 | 21.8 | 36.4 | 27.3 | 9.1
  > 0% reduction (T+M) | 62.1 | 65.2 | 78.2 | 63.6 | 72.7 | 90.9
  >= 25% reduction (T+M) | 31.0 | 47.2 | 51.7 | 36.4 | 36.4 | 63.6
  >= 50% reduction (T+M) | 10.3 | 28.1 | 25.3 | 9.1 | 36.4 | 36.4
  >= 75% reduction (T+M) | 4.6 | 10.1 | 8.0 | 9.1 | 9.1 | 0
  100% reduction (T+M) | 1.1 | 1.1 | 0 | 0 | 0 | 0
  Near Seizure free (T+M) | 1.1 | 2.2 | 1.1 | 0 | 0 | 0
  Worsening or No Change (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Worsening or No Change (M) | 40.2 | 35.2 | 20.9 | 36.4 | 27.3 | 9.1
  > 0% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  > 0% reduction (M) | 59.8 | 64.8 | 79.1 | 63.6 | 72.7 | 90.9
  >= 25% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 25% reduction (M) | 33.3 | 46.6 | 53.5 | 36.4 | 36.4 | 72.7
  >= 50% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 50% reduction (M) | 12.6 | 31.8 | 31.4 | 9.1 | 36.4 | 36.4
  >= 75% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 75% reduction (M) | 3.4 | 11.4 | 14.0 | 9.1 | 9.1 | 9.1
  100% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  100% reduction (M) | 1.1 | 3.4 | 2.3 | 0 | 9.1 | 0
  Near Seizure free (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Near Seizure free (M) | 1.1 | 4.5 | 2.3 | 9.1 | 9.1 | 0

18. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a Worsening From Baseline, or >0%, >=25%, >=50%, >=75%, 100% Reduction, and "Near Seizure Freedom" Between Baseline and T+M, and Baseline and M, in Seizures That Typically Results in Drops
Description: Seizures that typically result in drops included all: GTC, SGTC, TS, AS, and TA, whether confirmed by the ESC or not. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during T+M); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during combined T+M Period and Maintenance Period were reported.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percentage of participants
  Worsening or No Change (T+M) | 35.6 | 36.0 | 20.7 | 36.4 | 27.3 | 9.1
  > 0% reduction (T+M) | 64.4 | 64.0 | 79.3 | 63.6 | 72.7 | 90.9
  >= 25% reduction (T+M) | 31.0 | 46.1 | 50.6 | 36.4 | 36.4 | 63.6
  >= 50% reduction (T+M) | 9.2 | 27.0 | 26.4 | 9.1 | 36.4 | 36.4
  >= 75% reduction (T+M) | 3.4 | 9.0 | 8.0 | 9.1 | 9.1 | 0
  100% reduction (T+M) | 1.1 | 1.1 | 0 | 0 | 0 | 0
  Near Seizure free (T+M) | 1.1 | 1.1 | 1.1 | 0 | 0 | 0
  Worsening or No Change (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Worsening or No Change (M) | 37.9 | 37.5 | 19.8 | 36.4 | 27.3 | 9.1
  > 0% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  > 0% reduction (M) | 62.1 | 62.5 | 80.2 | 63.6 | 72.7 | 90.9
  >= 25% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 25% reduction (M) | 33.3 | 45.5 | 52.3 | 36.4 | 36.4 | 72.7
  >= 50% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 50% reduction (M) | 10.3 | 30.7 | 31.4 | 9.1 | 36.4 | 36.4
  >= 75% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 75% reduction (M) | 2.3 | 10.2 | 12.8 | 9.1 | 9.1 | 9.1
  100% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  100% reduction (M) | 1.1 | 2.3 | 2.3 | 0 | 9.1 | 0
  Near Seizure free (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Near Seizure free (M) | 1.1 | 2.3 | 2.3 | 9.1 | 9.1 | 0

19. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a Worsening From Baseline, or >0%, >=25%, >=50%, >=75%, 100% Reduction, and "Near Seizure Freedom" Between Baseline and T+M, and Baseline and M, in All Countable Motor Seizures
Description: Countable motor seizures included: GTC, SGTC, TS, AS, TA, CS, HS, and FS with clearly observable signs. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during T+M); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during combined T+M Period and Maintenance Period were reported.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percentage of participants
  Worsening or No Change (T+M) | 34.5 | 38.2 | 20.7 | 36.4 | 27.3 | 9.1
  > 0% reduction (T+M) | 65.5 | 61.8 | 79.3 | 63.6 | 72.7 | 90.9
  >= 25% reduction (T+M) | 33.3 | 44.9 | 50.6 | 36.4 | 36.4 | 63.6
  >= 50% reduction (T+M) | 9.2 | 24.7 | 25.3 | 9.1 | 36.4 | 36.4
  >= 75% reduction (T+M) | 2.3 | 9.0 | 6.9 | 9.1 | 9.1 | 0
  100% reduction (T+M) | 0 | 1.1 | 0 | 0 | 0 | 0
  Near Seizure free (T+M) | 0 | 1.1 | 0 | 0 | 0 | 0
  Worsening or No Change (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Worsening or No Change (M) | 36.8 | 38.6 | 18.6 | 36.4 | 27.3 | 9.1
  > 0% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  > 0% reduction (M) | 63.2 | 61.4 | 81.4 | 63.6 | 72.7 | 90.9
  >= 25% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 25% reduction (M) | 34.5 | 45.5 | 53.5 | 36.4 | 36.4 | 72.7
  >= 50% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 50% reduction (M) | 10.3 | 28.4 | 26.7 | 9.1 | 36.4 | 36.4
  >= 75% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 75% reduction (M) | 1.1 | 11.4 | 10.5 | 9.1 | 9.1 | 9.1
  100% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  100% reduction (M) | 0 | 2.3 | 1.2 | 0 | 9.1 | 0
  Near Seizure free (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Near Seizure free (M) | 0 | 2.3 | 1.2 | 9.1 | 9.1 | 0

20. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a Worsening From Baseline, or >0%, >=25%, >=50%, >=75%, 100% Reduction, and "Near Seizure Freedom" Between Baseline and T+M, and Baseline and M, in Countable Motor Seizures That do Not Result in Drops
Description: Countable motor seizures included: GTC, SGTC; TS, AS, TA, CS, HS, FS with clearly observable signs. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during T+M); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during combined T+M Period and Maintenance Period were reported.
Time Frame: as for outcome 17
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available. Here, number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed included those participants who were evaluable at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 70 | 73 | 64 | 8 | 7 | 9
percentage of participants
  Worsening or No Change (T+M) | 35.7 | 34.2 | 34.4 | 25.0 | 57.1 | 44.4
  > 0% reduction (T+M) | 64.3 | 65.8 | 65.6 | 75.0 | 42.9 | 55.6
  >= 25% reduction (T+M) | 51.4 | 53.4 | 46.9 | 50.0 | 14.3 | 44.4
  >= 50% reduction (T+M) | 30.0 | 43.8 | 32.8 | 25.0 | 0 | 22.2
  >= 75% reduction (T+M) | 12.9 | 26.0 | 12.5 | 12.5 | 0 | 11.1
  100% reduction (T+M) | 2.9 | 5.5 | 4.7 | 0 | 0 | 0
  Near Seizure free (T+M) | 2.9 | 9.6 | 7.8 | 0 | 0 | 0
  Worsening or No Change (M): number analyzed (Participants) | 70 | 72 | 63 | 8 | 7 | 9
  Worsening or No Change (M) | 31.4 | 33.3 | 34.9 | 25.0 | 57.1 | 44.4
  > 0% reduction (M): number analyzed (Participants) | 70 | 72 | 63 | 8 | 7 | 9
  > 0% reduction (M) | 68.6 | 66.7 | 65.1 | 75.0 | 42.9 | 55.6
  >= 25% reduction (M): number analyzed (Participants) | 70 | 72 | 63 | 8 | 7 | 9
  >= 25% reduction (M) | 54.3 | 56.9 | 49.2 | 50.0 | 14.3 | 44.4
  >= 50% reduction (M): number analyzed (Participants) | 70 | 72 | 63 | 8 | 7 | 9
  >= 50% reduction (M) | 31.4 | 44.4 | 33.3 | 25.0 | 0 | 22.2
  >= 75% reduction (M): number analyzed (Participants) | 70 | 72 | 63 | 8 | 7 | 9
  >= 75% reduction (M) | 17.1 | 29.2 | 17.5 | 12.5 | 0 | 11.1
  100% reduction (M): number analyzed (Participants) | 70 | 72 | 63 | 8 | 7 | 9
  100% reduction (M) | 5.7 | 9.7 | 6.3 | 12.5 | 0 | 0
  Near Seizure free (M): number analyzed (Participants) | 70 | 72 | 63 | 8 | 7 | 9
  Near Seizure free (M) | 7.1 | 13.9 | 9.5 | 12.5 | 0 | 0

21. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a Worsening From Baseline (ie <= 0% Reduction), or >0%, >=25%, >=50%, >=75%, 100% Reduction, and "Near Seizure Freedom" Between Baseline and T+M, and Baseline and M, in All Countable Seizures
Description: Countable motor seizures included: GTC, SGTC; TS, AS, TA, CS, HS, and FS with clearly observable signs. Countable non-motor seizures included: FS without clear observable signs, MS, absence/atypical absence, infantile spasms, epileptic spasms, and other seizures. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during T+M); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during combined T+M Period and Maintenance Period were reported.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percentage of participants
  Worsening or No Change (T+M) | 36.8 | 32.6 | 28.7 | 27.3 | 27.3 | 36.4
  > 0% reduction (T+M) | 63.2 | 67.4 | 71.3 | 72.7 | 72.7 | 63.6
  >= 25% reduction (T+M) | 35.6 | 48.3 | 46.0 | 27.3 | 27.3 | 45.5
  >= 50% reduction (T+M) | 11.5 | 22.5 | 20.7 | 9.1 | 27.3 | 27.3
  >= 75% reduction (T+M) | 3.4 | 6.7 | 4.6 | 9.1 | 9.1 | 0
  100% reduction (T+M) | 0 | 1.1 | 0 | 0 | 0 | 0
  Near Seizure free (T+M) | 0 | 1.1 | 0 | 0 | 0 | 0
  Worsening or No Change (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Worsening or No Change (M) | 34.5 | 33.0 | 27.9 | 27.3 | 27.3 | 27.3
  > 0% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  > 0% reduction (M) | 65.5 | 67.0 | 72.1 | 72.7 | 72.7 | 72.7
  >= 25% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 25% reduction (M) | 34.5 | 51.1 | 47.7 | 27.3 | 27.3 | 45.5
  >= 50% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 50% reduction (M) | 13.8 | 28.4 | 24.4 | 9.1 | 27.3 | 27.3
  >= 75% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  >= 75% reduction (M) | 3.4 | 9.1 | 7.0 | 9.1 | 9.1 | 0
  100% reduction (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  100% reduction (M) | 0 | 1.1 | 1.2 | 0 | 0 | 0
  Near Seizure free (M): number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  Near Seizure free (M) | 0 | 1.1 | 1.2 | 9.1 | 0 | 0

22. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a Worsening From Baseline, or >0%, >=25%, >=50%, >=75%, 100% Reduction, and "Near Seizure Freedom" Between Baseline and T+M, and Baseline and M, in All Countable Non-motor Seizures
Description: Countable non-motor seizures include: FS without clear observable signs, MS, absence/atypical absence, infantile spasms, epileptic spasms, and other seizures. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during T+M); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during combined T+M Period and Maintenance Period were reported.
Time Frame: as for outcome 17
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 63 | 64 | 57 | 8 | 7 | 8
percentage of participants
  Worsening or No Change (T+M) | 33.3 | 34.4 | 36.8 | 25.0 | 57.1 | 37.5
  > 0% reduction (T+M) | 66.7 | 65.6 | 63.2 | 75.0 | 42.9 | 62.5
  >= 25% reduction (T+M) | 52.4 | 56.3 | 43.9 | 50.0 | 14.3 | 37.5
  >= 50% reduction (T+M) | 30.2 | 48.4 | 35.1 | 25.0 | 0 | 25.0
  >= 75% reduction (T+M) | 14.3 | 32.8 | 12.3 | 12.5 | 0 | 0
  100% reduction (T+M) | 3.2 | 6.3 | 3.5 | 0 | 0 | 0
  Near Seizure free (T+M) | 3.2 | 14.1 | 5.3 | 0 | 0 | 0
  Worsening or No Change (M): number analyzed (Participants) | 63 | 63 | 56 | 8 | 7 | 8
  Worsening or No Change (M) | 30.2 | 30.2 | 33.9 | 12.5 | 57.1 | 37.5
  > 0% reduction (M): number analyzed (Participants) | 63 | 63 | 56 | 8 | 7 | 8
  > 0% reduction (M) | 69.8 | 69.8 | 66.1 | 87.5 | 42.9 | 62.5
  >= 25% reduction (M): number analyzed (Participants) | 63 | 63 | 56 | 8 | 7 | 8
  >= 25% reduction (M) | 54.0 | 60.3 | 48.2 | 50.0 | 14.3 | 37.5
  >= 50% reduction (M): number analyzed (Participants) | 63 | 63 | 56 | 8 | 7 | 8
  >= 50% reduction (M) | 34.9 | 49.2 | 33.9 | 25.0 | 0 | 37.5
  >= 75% reduction (M): number analyzed (Participants) | 63 | 63 | 56 | 8 | 7 | 8
  >= 75% reduction (M) | 17.5 | 31.7 | 17.9 | 12.5 | 0 | 0
  100% reduction (M): number analyzed (Participants) | 63 | 63 | 56 | 8 | 7 | 8
  100% reduction (M) | 6.3 | 9.5 | 8.9 | 12.5 | 0 | 0
  Near Seizure free (M): number analyzed (Participants) | 63 | 63 | 56 | 8 | 7 | 8
  Near Seizure free (M) | 7.9 | 15.9 | 10.7 | 12.5 | 0 | 0

23. Secondary Outcome: Part 1: Change From Baseline in Number of Seizure-free Days During T+M and M Period
Description: A day with no seizures leading to a drop was defined as a day for which electronic (e) diary data were available and no drop seizures were reported. The total number of drop seizure-free days was calculated per 28 days for Baseline and for T+M.
Time Frame: as for outcome 17
Population: The mITT population included all randomized participants who received at least 1 dose of ZX008 or placebo and for whom at least 1 week of diary data were available. Here, number analyzed included those participants who were evaluable for specified category.
Measure: Median (Full Range); unit: seizure free days per 28 days
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
seizure free days per 28 days
  T+M Period | 0.27 [-5.0 to 16.0] | 0.00 [-9.0 to 16.8] | 0.29 [-6.1 to 20.0] | 0.00 [-2.2 to 23.6] | 0.38 [-2.3 to 22.0] | 6.65 [-2.4 to 8.5]
  M Period: number analyzed (Participants) | 87 | 88 | 86 | 11 | 11 | 11
  M Period | 0.31 [-5.4 to 15.7] | 0.00 [-4.1 to 18.2] | 0.16 [-7.4 to 21.7] | -0.65 [-2.7 to 24.7] | 0.33 [-7.3 to 26.0] | 7.72 [-2.3 to 10.3]

24. Secondary Outcome: Part 1: Duration of Longest Interval (Days) Between Seizures That Result in Drops Comparing the ZX008 0.8 mg/kg/Day and 0.2 mg/kg/Day Groups Independently Versus Placebo
Description: The longest interval between seizures leading to drops were obtained from the eDiary entries in Titration and Maintenance Period. The interval was derived as the maximum value of the number of days between consecutive drop seizures.
Time Frame: From Baseline up to 14 weeks [Titration Period (2 weeks) + Maintenance Period (12 weeks)]
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
days | 5.00 [1.0 to 39.0] | 4.00 [1.0 to 97.0] | 5.00 [1.0 to 89.0] | 4.00 [1.0 to 91.0] | 4.00 [1.0 to 32.0] | 6.00 [2.0 to 16.0]

25. Secondary Outcome: Part 1: Clinical Global Impression - Improvement as Assessed by the Parent/Caregiver
Description: CGI-I scale measures improvement in the participant's condition from Baseline. The severity of a participant's condition was rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), as follows: 1-very much improved, 2-much improved, 3-minimally improved, 4- no change, 5-minimally worse, 6-much worse and 7-very much worse.
Time Frame: At Days 15, 43, 71 and 99
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 85 | 85 | 81 | 11 | 11 | 11
percentage of participants
  1=Very much improved (D15): number analyzed (Participants) | 85 | 85 | 81 | 11 | 10 | 11
  1=Very much improved (D15) | 2.4 | 5.9 | 9.9 | 9.1 | 10.0 | 9.1
  2=Much improved (D15): number analyzed (Participants) | 85 | 85 | 81 | 11 | 10 | 11
  2=Much improved (D15) | 4.7 | 15.3 | 21.0 | 18.2 | 10.0 | 18.2
  3=Minimally improved (D15): number analyzed (Participants) | 85 | 85 | 81 | 11 | 10 | 11
  3=Minimally improved (D15) | 31.8 | 27.1 | 39.5 | 9.1 | 30.0 | 27.3
  4=No Change (D15): number analyzed (Participants) | 85 | 85 | 81 | 11 | 10 | 11
  4=No Change (D15) | 51.8 | 42.4 | 18.5 | 63.6 | 30.0 | 27.3
  5=Minimally worse (D15): number analyzed (Participants) | 85 | 85 | 81 | 11 | 10 | 11
  5=Minimally worse (D15) | 4.7 | 5.9 | 7.4 | 0 | 20.0 | 18.2
  6=Much worse (D15): number analyzed (Participants) | 85 | 85 | 81 | 11 | 10 | 11
  6=Much worse (D15) | 4.7 | 3.5 | 2.5 | 0 | 0 | 0
  7=Very much worse (D15): number analyzed (Participants) | 85 | 85 | 81 | 11 | 10 | 11
  7=Very much worse (D15) | 0 | 0 | 1.2 | 0 | 0 | 0
  1=Very much improved (D43): number analyzed (Participants) | 85 | 82 | 80 | 11 | 9 | 10
  1=Very much improved (D43) | 1.2 | 7.3 | 13.8 | 9.1 | 0 | 10.0
  2=Much improved (D43): number analyzed (Participants) | 85 | 82 | 80 | 11 | 9 | 10
  2=Much improved (D43) | 9.4 | 19.5 | 25.0 | 0 | 22.2 | 40.0
  3=Minimally improved (D43): number analyzed (Participants) | 85 | 82 | 80 | 11 | 9 | 10
  3=Minimally improved (D43) | 20.0 | 18.3 | 33.8 | 18.2 | 44.4 | 30.0
  4=No Change (D43): number analyzed (Participants) | 85 | 82 | 80 | 11 | 9 | 10
  4=No Change (D43) | 60.0 | 39.0 | 17.5 | 63.6 | 33.3 | 0
  5=Minimally worse (D43): number analyzed (Participants) | 85 | 82 | 80 | 11 | 9 | 10
  5=Minimally worse (D43) | 5.9 | 11.0 | 5.0 | 9.1 | 0 | 20.0
  6=Much worse (D43): number analyzed (Participants) | 85 | 82 | 80 | 11 | 9 | 10
  6=Much worse (D43) | 2.4 | 4.9 | 5.0 | 0 | 0 | 0
  7=Very much worse (D43): number analyzed (Participants) | 85 | 82 | 80 | 11 | 9 | 10
  7=Very much worse (D43) | 1.2 | 0 | 0 | 0 | 0 | 0
  1=Very much improved (D71): number analyzed (Participants) | 82 | 75 | 75 | 11 | 9 | 9
  1=Very much improved (D71) | 2.4 | 4.0 | 10.7 | 9.1 | 0 | 0
  2=Much improved (D71): number analyzed (Participants) | 82 | 75 | 75 | 11 | 9 | 9
  2=Much improved (D71) | 6.1 | 20.0 | 28.0 | 0 | 22.2 | 11.1
  3=Minimally improved (D71): number analyzed (Participants) | 82 | 75 | 75 | 11 | 9 | 9
  3=Minimally improved (D71) | 24.4 | 16.0 | 33.3 | 18.2 | 22.2 | 55.6
  4=No Change (D71): number analyzed (Participants) | 82 | 75 | 75 | 11 | 9 | 9
  4=No Change (D71) | 53.7 | 48.0 | 24.0 | 63.6 | 55.6 | 22.2
  5=Minimally worse (D71): number analyzed (Participants) | 82 | 75 | 75 | 11 | 9 | 9
  5=Minimally worse (D71) | 7.3 | 8.0 | 1.3 | 9.1 | 0 | 11.1
  6=Much worse (D71): number analyzed (Participants) | 82 | 75 | 75 | 11 | 9 | 9
  6=Much worse (D71) | 6.1 | 4.0 | 2.7 | 0 | 0 | 0
  7=Very much worse (D71): number analyzed (Participants) | 82 | 75 | 75 | 11 | 9 | 9
  7=Very much worse (D71) | 0 | 0 | 0 | 0 | 0 | 0
  1=Very much improved (D99): number analyzed (Participants) | 81 | 85 | 80 | 11 | 11 | 11
  1=Very much improved (D99) | 1.2 | 8.2 | 10.0 | 9.1 | 0 | 18.2
  2=Much improved (D99): number analyzed (Participants) | 81 | 85 | 80 | 11 | 11 | 11
  2=Much improved (D99) | 3.7 | 18.8 | 23.8 | 0 | 18.2 | 18.2
  3=Minimally improved (D99): number analyzed (Participants) | 81 | 85 | 80 | 11 | 11 | 11
  3=Minimally improved (D99) | 32.1 | 16.5 | 27.5 | 18.2 | 27.3 | 36.4
  4=No Change (D99): number analyzed (Participants) | 81 | 85 | 80 | 11 | 11 | 11
  4=No Change (D99) | 53.1 | 37.6 | 27.5 | 63.6 | 45.5 | 27.3
  5=Minimally worse (D99): number analyzed (Participants) | 81 | 85 | 80 | 11 | 11 | 11
  5=Minimally worse (D99) | 7.4 | 8.2 | 5.0 | 0 | 9.1 | 0
  6=Much worse (D99): number analyzed (Participants) | 81 | 85 | 80 | 11 | 11 | 11
  6=Much worse (D99) | 2.5 | 7.1 | 5.0 | 9.1 | 0 | 0
  7=Very much worse (D99): number analyzed (Participants) | 81 | 85 | 80 | 11 | 11 | 11
  7=Very much worse (D99) | 0 | 3.5 | 1.3 | 0 | 0 | 0

26. Secondary Outcome: Part 1: Percentage of Participants With TEAEs
Description: Adverse events were defined as any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A TEAE in Part 1 was defined as any AE that, based on start date information, occurred after the first dose of study drug in Part 1, but not on or after the first dose of study drug in Part 2.
Time Frame: Baseline up to 14 weeks + Taper/Transition (2 weeks)
Population: The Safety Population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percentage of participants | 80.5 | 78.7 | 89.7 | 72.7 | 90.9 | 63.6

27. Secondary Outcome: Part 1: Percentage of Participants With Serious TEAEs
Description: as for outcome 3
Time Frame: Baseline up to 14 weeks + Taper/Transition (2 weeks)
Population: The Safety Population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Placebo | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day | Cohort B: Placebo | Cohort B: ZX008 0.2 mg/kg/Day | Cohort B: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 87 | 89 | 87 | 11 | 11 | 11
percentage of participants | 4.6 | 4.5 | 11.5 | 9.1 | 9.1 | 0

28. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration of Fenfluramine and Norfenfluramine Determined Directly From the Concentration Time Profile [Cmax] at Steady State
Description: Cmax is the maximum plasma concentration determined directly from the concentration time profile.
Time Frame: At Visit 8 (Day 43) of the Maintenance Period: pre-dose, 1, 2, and 4-6 hours post-dose
Population: The Pharmacokinetic (PK) analysis set included those participants who received at least one dose of ZX008 and at least one plasma concentration measurement in Study ZX008-1601.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 84 | 80
nanograms per milliliter (ng/mL)
  Fenfluramine | 11.9 (56.1) | 44.8 (47.0)
  Norfenfluramine | 9.04 (53.4) | 28.9 (52.9)

29. Secondary Outcome: Part 1: Minimum Observed Plasma Concentration of Fenfluramine and Norfenfluramine at Steady State Determined Directly From the Concentration-time Profile [Cmin] at Steady State
Description: Cmin is the minimum plasma concentration determined directly from the concentration-time profile.
Time Frame: At Visit 8 (Day 43) of the Maintenance Period: pre-dose, 1, 2, and 4-6 hours post-dose
Population: The PK analysis set included those participants who received at least one dose of ZX008 and at least one plasma concentration measurement in Study ZX008-1601.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 84 | 80
ng/mL
  Fenfluramine | 8.19 (75.6) | 31.8 (60.8)
  Norfenfluramine | 8.23 (61.3) | 26.2 (58.9)

30. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of Fenfluramine and Norfenfluramine From Time Zero to Time 24 Hours [AUC0-24hours] at Steady State
Description: AUC0-24 is the area under the concentration-time curve from time 0 to 24 hours.
Time Frame: At Visit 8 (Day 43) of the Maintenance Period: pre-dose, 1, 2, and 4-6 hours post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Cohort A: ZX008 0.2 mg/kg/Day | Cohort A: ZX008 0.8 mg/kg/Day
Number analyzed (Participants) | 84 | 80
nanograms*hour per milliliter (ng*h/mL)
  Fenfluramine | 246 (63.0) | 933 (52.1)
  Norfenfluramine | 209 (56.3) | 667 (55.1)

31. Secondary Outcome: Part 2: Percent Change From Baseline in the Frequency of Seizures That Result in Drops (ESC Confirmed) in OLE Period
Description: as for outcome 11
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: The Open-Label Extension Modified Intent-To-Treat (mITT) Population included all participants who received at least 1 dose of ZX008 and had a valid estimate of the frequency of seizures that resulted in drops from Part 1 and at least 1 month (30 days) of valid seizure data during the OLE. As pre-specified in study design, participants in Part 2 received individualized optimized treatment (0.2 mg/kg/day to 0.8 mg/kg/day) based on Investigator discretion. Hence overall data for Part 2 is reported.
Measure: Median (Full Range); unit: percent change
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percent change | -29.53 [-100.0 to 2625.3] | -43.42 [-99.0 to 64.2]

32. Secondary Outcome: Part 2: Percent Change From Baseline in the Frequency of All Seizures That Typically Result in Drops Between Baseline and the OLE Period Whether ESC Confirmed as Drop or Not
Description: as for outcome 7
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: The OLE mITT population included all participants who received at least 1 dose of ZX008 and had a valid estimate of the frequency of seizures that resulted in drops from Part 1 and at least 1 month (30 days) of valid seizure data during the OLE. As pre-specified in study design, participants in Part 2 received individualized optimized treatment (0.2 mg/kg/day to 0.8 mg/kg/day) based on Investigator discretion. Hence overall data for Part 2 is reported.
Measure: Median (Full Range); unit: percent change
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percent change | -27.94 [-100.0 to 2625.3] | -43.78 [-99.0 to 64.2]

33. Secondary Outcome: Part 2: Percent Change From Baseline in the Frequency of All Countable Motor Seizures in OLE Period
Description: as for outcome 8
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percent change | -28.18 [-100.0 to 2625.3] | -41.94 [-99.0 to 64.2]

34. Secondary Outcome: Part 2: Change From Baseline in the Frequency of All Countable Non-motor Seizures in OLE Period
Description: as for outcome 9
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
seizure frequency per 28 days | 0.00 [-4257.2 to 1774.3] | 0.00 [-89.4 to 258.9]

35. Secondary Outcome: Part 2: Percent Change From Baseline in the Frequency of All Countable Seizures (ESC Confirmed or Not) in OLE Period
Description: as for outcome 10
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Median (Full Range); unit: percent change
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percent change | -28.83 [-100.0 to 606.1] | -28.00 [-99.1 to 83.3]

36. Secondary Outcome: Part 2: Change From Baseline in the Frequency of All Countable Seizures That Did Not Result in Drops (ESC Confirmed) in OLE Period
Description: Nondrop seizures were defined as any countable seizure types that did not meet the criteria of drop seizures, ie, are classified as CS, HC, FS with or without observable signs, MS, absence/atypical absence, infantile spasms, epileptic spasms, or other; or are seizures of the following classifications that were approved for each subject as non-drop seizure types by the ESC: GTC, SGTC, TS, AS, or TA. For each participant, the seizure frequency per 28 days was calculated as the number of seizures recorded during the period, divided by the number of days in the period and multiplied by 28.
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
seizure frequency per 28 days | -0.99 [-4482.2 to 1774.3] | 0.00 [-89.4 to 258.9]

37. Secondary Outcome: Part 2: Percentage of Participants Who Achieved a Worsening From Baseline, or > 0%, >=25%, >= 50%, >= 75%, 100% Reduction, and "Near Seizure Freedom" From Baseline in Frequency of Seizures That Result in Drops (ESC Confirmed)
Description: The seizure types included in the count were: atonic, tonic, tonic/atonic, generalized tonic-clonic, and secondarily generalized tonic-clonic seizures resulting in drops. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during OLE Period); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during OLE Period were reported.
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percentage of participants
  Worsening or No Change | 31.5 | 18.8
  > 0% | 68.5 | 81.3
  >= 25% | 55.6 | 62.5
  >= 50% | 32.8 | 43.8
  >= 75% | 12.4 | 21.9
  100% | 1.2 | 0
  Near Seizure free | 1.7 | 0

38. Secondary Outcome: Part 2: Percentage of Participants Who Achieved a Worsening From Baseline, or > 0%, >=25%, >= 50%, >= 75%, 100% Reduction, and "Near Seizure Freedom" From Baseline in Frequency of Seizures That Typically Result in Drops
Description: Seizures that typically result in drops included all: GTC, SGTC, TS, AS, and TA, whether confirmed by the ESC or not. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during OLE Period); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during OLE Period were reported.
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percentage of participants
  Worsening or No Change | 32.0 | 21.9
  > 0% | 68.0 | 78.1
  >= 25% | 53.1 | 65.6
  >= 50% | 29.9 | 43.8
  >= 75% | 11.2 | 21.9
  100% | 0.8 | 0
  Near Seizure free | 1.2 | 0

39. Secondary Outcome: Part 2: Percentage of Participants Who Achieved a Worsening From Baseline, or > 0%, >=25%, >= 50%, >= 75%, 100% Reduction, and "Near Seizure Freedom" From Baseline in Frequency of All Countable Motor Seizures
Description: Countable motor seizures included: GTC, SGTC, TS, AS, TA, CS, HS, and FS with clearly observable signs. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during OLE Period); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during OLE Period were reported.
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percentage of participants
  Worsening or No Change | 29.5 | 21.9
  > 0% | 70.5 | 78.1
  >= 25% | 54.8 | 62.5
  >= 50% | 29.9 | 40.6
  >= 75% | 9.1 | 21.9
  100% | 0.4 | 0
  Near Seizure free | 0.8 | 0

40. Secondary Outcome: Part 2: Percentage of Participants Who Achieved a Worsening From Baseline, or > 0%, >=25%, >= 50%, >= 75%, 100% Reduction, and "Near Seizure Freedom" From Baseline in Frequency of All Countable Non-motor Seizures
Description: Countable non-motor seizures included: FS without clear observable signs, MS, absence/atypical absence, infantile spasms, epileptic spasms, and other seizures. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during OLE Period); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during OLE Period were reported.
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percentage of participants
  Worsening or No Change | 24.1 | 37.5
  > 0% | 46.1 | 31.3
  >= 25% | 41.9 | 25.0
  >= 50% | 34.0 | 18.8
  >= 75% | 22.8 | 6.3
  100% | 4.6 | 3.1
  Near Seizure free | 7.5 | 6.3

41. Secondary Outcome: Part 2: Percentage of Participants Who Achieved a Worsening From Baseline, or > 0%, >=25%, >= 50%, >= 75%, 100% Reduction, and "Near Seizure Freedom" From Baseline in Frequency of All Countable Seizures
Description: Countable motor seizures included: GTC, SGTC; TS, AS, TA, CS, HS, and FS with clearly observable signs. Countable non-motor seizures included: FS without clear observable signs, MS, absence/atypical absence, infantile spasms, epileptic spasms, and other seizures. The participants who experienced a worsening or no change from Baseline (ie <= 0% reduction); >0%, >=25%, >=50%, >=75%, and 100% reduction (a 100% reduction was equivalent to achieving seizure freedom during OLE Period); and "near seizure freedom," (defined as 0 or 1 seizure leading to a drop) during OLE Period were reported.
Time Frame: From OLE Month 1 to Month12, compared to Baseline (Part 1)
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
percentage of participants
  Worsening or No Change | 30.3 | 37.5
  > 0% | 69.7 | 62.5
  >= 25% | 53.1 | 56.3
  >= 50% | 30.7 | 28.1
  >= 75% | 9.1 | 12.5
  100% | 0.4 | 0
  Near Seizure free | 0.4 | 0

42. Secondary Outcome: Part 2: Change From Baseline in Number of Seizure-free Days Per 28 Days (ESC Confirmed) in OLE Period
Description: A day with no seizures leading to a drop was defined as a day for which ediary data were available and no drop seizures were reported.
Time Frame: From Part 2 Baseline until end of OLE Period (up to 72 months)
Population: as for outcome 32
Measure: Median (Full Range); unit: seizure free days per 28 days
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 32
seizure free days per 28 days | 2.16 [-23.0 to 27.8] | 4.24 [-3.6 to 24.5]

43. Secondary Outcome: Part 2: Change From Baseline in Duration of Longest Interval Between Seizures That Result in Drops (ESC Confirmed) in OLE Period
Description: The longest interval between seizures leading to drops were obtained from the eDiary entries in OLE Period. The interval was derived as the maximum value of the number of days between consecutive drop seizures.
Time Frame: From Part 2 Baseline until end of the OLE Period (up to 72 months)
Population: OLE mITT:all participants who received at least 1 dose of ZX008 and had valid estimate of frequency of seizures that resulted in drops from Part 1 and at least 1 month(30 days) of valid seizure data during OLE. Number of participants analyzed=participants who were evaluable for assessment. As pre-specified in study design, participants in Part 2 received individualized optimized treatment(0.2 mg/kg/day to 0.8 mg/kg/day) based on Investigator discretion. Hence overall data for Part 2 is reported.
Measure: Median (Full Range); unit: days
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 241 | 27
days | 4.0 [-10 to 360] | 6.0 [0 to 200]

44. Secondary Outcome: Part 2: Clinical Global Impression - Improvement as Assessed by the Principal Investigator
Description: CGI-I scale measures improvement in the participant's condition from Baseline. The severity of a participant's condition was rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), as follows: 1-very much improved,2-much improved, 3-minimally improved, 4- no change, 5-minimally worse, 6-much worse and 7-very much worse.
Time Frame: At OLE Day 1, OLE Months (M) 1, 2, 3, 6, 9, 12, and Last Assessment (up to 72 months)
Population: OLE mITT:participants who received >=1 dose of ZX008, had valid estimate of frequency of seizures that resulted in drops from Part 1 and at least 1 month(30 days) of valid seizure data during OLE. N: participants evaluable for assessment. n: participants evaluable at specified time point. As pre-specified in study design, participants in Part 2 received individualized optimized treatment (0.2 mg/kg/day to 0.8 mg/kg/day) based on Investigator discretion. Hence overall data for Part 2 is reported.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 237 | 32
percentage of participants
  1=Very much improved (OLE D1): number analyzed (Participants) | 236 | 32
  1=Very much improved (OLE D1) | 2.5 | 3.1
  2=Much improved (OLE D1): number analyzed (Participants) | 236 | 32
  2=Much improved (OLE D1) | 15.3 | 18.8
  3=Minimally improved (OLE D1): number analyzed (Participants) | 236 | 32
  3=Minimally improved (OLE D1) | 25.8 | 18.8
  4=No Change (OLE D1): number analyzed (Participants) | 236 | 32
  4=No Change (OLE D1) | 48.3 | 56.3
  5=Minimally worse (OLE D1): number analyzed (Participants) | 236 | 32
  5=Minimally worse (OLE D1) | 7.2 | 3.1
  6=Much worse (OLE D1): number analyzed (Participants) | 236 | 32
  6=Much worse (OLE D1) | 0.8 | 0
  7=Very much worse (OLE D1): number analyzed (Participants) | 236 | 32
  7=Very much worse (OLE D1) | 0 | 0
  1=Very much improved (OLE M1): number analyzed (Participants) | 225 | 32
  1=Very much improved (OLE M1) | 4.4 | 9.4
  2=Much improved (OLE M1): number analyzed (Participants) | 225 | 32
  2=Much improved (OLE M1) | 20.0 | 21.9
  3=Minimally improved (OLE M1): number analyzed (Participants) | 225 | 32
  3=Minimally improved (OLE M1) | 32.4 | 37.5
  4=No Change (OLE M1): number analyzed (Participants) | 225 | 32
  4=No Change (OLE M1) | 34.2 | 31.3
  5=Minimally worse (OLE M1): number analyzed (Participants) | 225 | 32
  5=Minimally worse (OLE M1) | 7.6 | 0
  6=Much worse (OLE M1): number analyzed (Participants) | 225 | 32
  6=Much worse (OLE M1) | 1.3 | 0
  7=Very much worse (OLE M1): number analyzed (Participants) | 225 | 32
  7=Very much worse (OLE M1) | 0 | 0
  1=Very much improved (OLE M2): number analyzed (Participants) | 220 | 31
  1=Very much improved (OLE M2) | 5.5 | 6.5
  2=Much improved (OLE M2): number analyzed (Participants) | 220 | 31
  2=Much improved (OLE M2) | 24.5 | 19.4
  3=Minimally improved (OLE M2): number analyzed (Participants) | 220 | 31
  3=Minimally improved (OLE M2) | 34.1 | 35.5
  4=No Change (OLE M2): number analyzed (Participants) | 220 | 31
  4=No Change (OLE M2) | 27.7 | 32.3
  5=Minimally worse (OLE M2): number analyzed (Participants) | 220 | 31
  5=Minimally worse (OLE M2) | 5.0 | 6.5
  6=Much worse (OLE M2): number analyzed (Participants) | 220 | 31
  6=Much worse (OLE M2) | 3.2 | 0
  7=Very much worse (OLE M2): number analyzed (Participants) | 220 | 31
  7=Very much worse (OLE M2) | 0 | 0
  1=Very much improved (OLE M3): number analyzed (Participants) | 207 | 29
  1=Very much improved (OLE M3) | 7.2 | 6.9
  2=Much improved (OLE M3): number analyzed (Participants) | 207 | 29
  2=Much improved (OLE M3) | 25.1 | 17.2
  3=Minimally improved (OLE M3): number analyzed (Participants) | 207 | 29
  3=Minimally improved (OLE M3) | 36.2 | 55.2
  4=No Change (OLE M3): number analyzed (Participants) | 207 | 29
  4=No Change (OLE M3) | 21.7 | 20.7
  5=Minimally worse (OLE M3): number analyzed (Participants) | 207 | 29
  5=Minimally worse (OLE M3) | 7.2 | 0
  6=Much worse (OLE M3): number analyzed (Participants) | 207 | 29
  6=Much worse (OLE M3) | 2.4 | 0
  7=Very much worse (OLE M3): number analyzed (Participants) | 207 | 29
  7=Very much worse (OLE M3) | 0 | 0
  1=Very much improved (OLE M6): number analyzed (Participants) | 184 | 29
  1=Very much improved (OLE M6) | 8.2 | 3.4
  2=Much improved (OLE M6): number analyzed (Participants) | 184 | 29
  2=Much improved (OLE M6) | 33.7 | 27.6
  3=Minimally improved (OLE M6): number analyzed (Participants) | 184 | 29
  3=Minimally improved (OLE M6) | 31.0 | 34.5
  4=No Change (OLE M6): number analyzed (Participants) | 184 | 29
  4=No Change (OLE M6) | 20.1 | 27.6
  5=Minimally worse (OLE M6): number analyzed (Participants) | 184 | 29
  5=Minimally worse (OLE M6) | 3.8 | 6.9
  6=Much worse (OLE M6): number analyzed (Participants) | 184 | 29
  6=Much worse (OLE M6) | 3.3 | 0
  7=Very much worse (OLE M6): number analyzed (Participants) | 184 | 29
  7=Very much worse (OLE M6) | 0 | 0
  1=Very much improved (OLE M9): number analyzed (Participants) | 133 | 28
  1=Very much improved (OLE M9) | 9.0 | 3.6
  2=Much improved (OLE M9): number analyzed (Participants) | 133 | 28
  2=Much improved (OLE M9) | 37.6 | 28.6
  3=Minimally improved (OLE M9): number analyzed (Participants) | 133 | 28
  3=Minimally improved (OLE M9) | 27.1 | 28.6
  4=No Change (OLE M9): number analyzed (Participants) | 133 | 28
  4=No Change (OLE M9) | 18.8 | 35.7
  5=Minimally worse (OLE M9): number analyzed (Participants) | 133 | 28
  5=Minimally worse (OLE M9) | 6.0 | 3.6
  6=Much worse (OLE M9): number analyzed (Participants) | 133 | 28
  6=Much worse (OLE M9) | 1.5 | 0
  7=Very much worse (OLE M9): number analyzed (Participants) | 133 | 28
  7=Very much worse (OLE M9) | 0 | 0
  1=Very much improved (OLE M12): number analyzed (Participants) | 145 | 26
  1=Very much improved (OLE M12) | 9.7 | 0
  2=Much improved (OLE M12): number analyzed (Participants) | 145 | 26
  2=Much improved (OLE M12) | 39.3 | 53.8
  3=Minimally improved (OLE M12): number analyzed (Participants) | 145 | 26
  3=Minimally improved (OLE M12) | 26.2 | 23.1
  4=No Change (OLE M12): number analyzed (Participants) | 145 | 26
  4=No Change (OLE M12) | 18.6 | 19.2
  5=Minimally worse (OLE M12): number analyzed (Participants) | 145 | 26
  5=Minimally worse (OLE M12) | 3.4 | 3.8
  6=Much worse (OLE M12): number analyzed (Participants) | 145 | 26
  6=Much worse (OLE M12) | 2.8 | 0
  7=Very much worse (OLE M12): number analyzed (Participants) | 145 | 26
  7=Very much worse (OLE M12) | 0 | 0
  1=Very much improved (Last Assessment) | 7.6 | 6.3
  2=Much improved (Last Assessment) | 27.4 | 25.0
  3=Minimally improved (Last Assessment) | 21.9 | 25.0
  4=No Change (Last Assessment) | 28.3 | 40.6
  5=Minimally worse (Last Assessment) | 7.2 | 3.1
  6=Much worse (Last Assessment) | 7.6 | 0
  7=Very much worse (Last Assessment) | 0 | 0

45. Secondary Outcome: Part 2: Clinical Global Impression - Improvement as Assessed by the Parent/Caregiver
Description: as for outcome 44
Time Frame: At OLE Day 1, OLE Months (M) 1, 2, 3, 6, 9, 12, and Last Assessment (up to 72 months)
Population: OLE mITT:all participants who received >= 1 dose of ZX008, had valid estimate of frequency of seizures that resulted in drops from Part 1 and >= 1 month(30 days) of valid seizure data during OLE. N: participants evaluable for assessment. n: participants evaluable at specified time point. As pre-specified in study design, participants in Part 2 received individualized optimized treatment (0.2 mg/kg/day to 0.8 mg/kg/day) based on Investigator discretion. Hence overall data for Part 2 is reported.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Cohort A- Overall | Part 2: Cohort B- Overall
Number analyzed (Participants) | 237 | 32
percentage of participants
  1=Very much improved (OLE D1): number analyzed (Participants) | 232 | 32
  1=Very much improved (OLE D1) | 6.9 | 9.4
  2=Much improved (OLE D1): number analyzed (Participants) | 232 | 32
  2=Much improved (OLE D1) | 16.8 | 12.5
  3=Minimally improved (OLE D1): number analyzed (Participants) | 232 | 32
  3=Minimally improved (OLE D1) | 24.6 | 28.1
  4=No Change (OLE D1): number analyzed (Participants) | 232 | 32
  4=No Change (OLE D1) | 40.1 | 43.8
  5=Minimally worse (OLE D1): number analyzed (Participants) | 232 | 32
  5=Minimally worse (OLE D1) | 6.9 | 3.1
  6=Much worse (OLE D1): number analyzed (Participants) | 232 | 32
  6=Much worse (OLE D1) | 3.9 | 3.1
  7=Very much worse (OLE D1): number analyzed (Participants) | 232 | 32
  7=Very much worse (OLE D1) | 0.9 | 0
  1=Very much improved (OLE M1): number analyzed (Participants) | 224 | 32
  1=Very much improved (OLE M1) | 7.1 | 12.5
  2=Much improved (OLE M1): number analyzed (Participants) | 224 | 32
  2=Much improved (OLE M1) | 21.4 | 15.6
  3=Minimally improved (OLE M1): number analyzed (Participants) | 224 | 32
  3=Minimally improved (OLE M1) | 32.1 | 31.3
  4=No Change (OLE M1): number analyzed (Participants) | 224 | 32
  4=No Change (OLE M1) | 29.5 | 40.6
  5=Minimally worse (OLE M1): number analyzed (Participants) | 224 | 32
  5=Minimally worse (OLE M1) | 5.8 | 0
  6=Much worse (OLE M1): number analyzed (Participants) | 224 | 32
  6=Much worse (OLE M1) | 4.0 | 0
  7=Very much worse (OLE M1): number analyzed (Participants) | 224 | 32
  7=Very much worse (OLE M1) | 0 | 0
  1=Very much improved (OLE M2): number analyzed (Participants) | 219 | 31
  1=Very much improved (OLE M2) | 7.3 | 12.9
  2=Much improved (OLE M2): number analyzed (Participants) | 219 | 31
  2=Much improved (OLE M2) | 25.6 | 16.1
  3=Minimally improved (OLE M2): number analyzed (Participants) | 219 | 31
  3=Minimally improved (OLE M2) | 32.0 | 41.9
  4=No Change (OLE M2): number analyzed (Participants) | 219 | 31
  4=No Change (OLE M2) | 25.6 | 22.6
  5=Minimally worse (OLE M2): number analyzed (Participants) | 219 | 31
  5=Minimally worse (OLE M2) | 6.4 | 6.5
  6=Much worse (OLE M2): number analyzed (Participants) | 219 | 31
  6=Much worse (OLE M2) | 2.3 | 0
  7=Very much worse (OLE M2): number analyzed (Participants) | 219 | 31
  7=Very much worse (OLE M2) | 0.9 | 0
  1=Very much improved (OLE M3): number analyzed (Participants) | 207 | 29
  1=Very much improved (OLE M3) | 9.7 | 13.8
  2=Much improved (OLE M3): number analyzed (Participants) | 207 | 29
  2=Much improved (OLE M3) | 30.0 | 10.3
  3=Minimally improved (OLE M3): number analyzed (Participants) | 207 | 29
  3=Minimally improved (OLE M3) | 29.5 | 37.9
  4=No Change (OLE M3): number analyzed (Participants) | 207 | 29
  4=No Change (OLE M3) | 19.3 | 37.9
  5=Minimally worse (OLE M3): number analyzed (Participants) | 207 | 29
  5=Minimally worse (OLE M3) | 9.7 | 0
  6=Much worse (OLE M3): number analyzed (Participants) | 207 | 29
  6=Much worse (OLE M3) | 0.5 | 0
  7=Very much worse (OLE M3): number analyzed (Participants) | 207 | 29
  7=Very much worse (OLE M3) | 1.4 | 0
  1=Very much improved (OLE M6): number analyzed (Participants) | 186 | 29
  1=Very much improved (OLE M6) | 13.4 | 10.3
  2=Much improved (OLE M6): number analyzed (Participants) | 186 | 29
  2=Much improved (OLE M6) | 30.1 | 31.0
  3=Minimally improved (OLE M6): number analyzed (Participants) | 186 | 29
  3=Minimally improved (OLE M6) | 27.4 | 34.5
  4=No Change (OLE M6): number analyzed (Participants) | 186 | 29
  4=No Change (OLE M6) | 23.1 | 20.7
  5=Minimally worse (OLE M6): number analyzed (Participants) | 186 | 29
  5=Minimally worse (OLE M6) | 3.2 | 0
  6=Much worse (OLE M6): number analyzed (Participants) | 186 | 29
  6=Much worse (OLE M6) | 2.2 | 3.4
  7=Very much worse (OLE M6): number analyzed (Participants) | 186 | 29
  7=Very much worse (OLE M6) | 0.5 | 0
  1=Very much improved (OLE M9): number analyzed (Participants) | 134 | 28
  1=Very much improved (OLE M9) | 13.4 | 14.3
  2=Much improved (OLE M9): number analyzed (Participants) | 134 | 28
  2=Much improved (OLE M9) | 37.3 | 25.0
  3=Minimally improved (OLE M9): number analyzed (Participants) | 134 | 28
  3=Minimally improved (OLE M9) | 26.1 | 21.4
  4=No Change (OLE M9): number analyzed (Participants) | 134 | 28
  4=No Change (OLE M9) | 14.2 | 32.1
  5=Minimally worse (OLE M9): number analyzed (Participants) | 134 | 28
  5=Minimally worse (OLE M9) | 8.2 | 3.6
  6=Much worse (OLE M9): number analyzed (Participants) | 134 | 28
  6=Much worse (OLE M9) | 0.7 | 3.6
  7=Very much worse (OLE M9): number analyzed (Participants) | 134 | 28
  7=Very much worse (OLE M9) | 0 | 0
  1=Very much improved (OLE M12): number analyzed (Participants) | 149 | 26
  1=Very much improved (OLE M12) | 16.8 | 19.2
  2=Much improved (OLE M12): number analyzed (Participants) | 149 | 26
  2=Much improved (OLE M12) | 34.2 | 26.9
  3=Minimally improved (OLE M12): number analyzed (Participants) | 149 | 26
  3=Minimally improved (OLE M12) | 26.8 | 46.2
  4=No Change (OLE M12): number analyzed (Participants) | 149 | 26
  4=No Change (OLE M12) | 14.8 | 3.8
  5=Minimally worse (OLE M12): number analyzed (Participants) | 149 | 26
  5=Minimally worse (OLE M12) | 4.7 | 3.8
  6=Much worse (OLE M12): number analyzed (Participants) | 149 | 26
  6=Much worse (OLE M12) | 2.0 | 0
  7=Very much worse (OLE M12): number analyzed (Participants) | 149 | 26
  7=Very much worse (OLE M12) | 0.7 | 0
  1=Very much improved (Last Assessment) | 11.4 | 12.5
  2=Much improved (Last Assessment) | 24.1 | 28.1
  3=Minimally improved (Last Assessment) | 24.5 | 18.8
  4=No Change (Last Assessment) | 25.3 | 28.1
  5=Minimally worse (Last Assessment) | 9.3 | 9.4
  6=Much worse (Last Assessment) | 3.4 | 3.1
  7=Very much worse (Last Assessment) | 2.1 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to 72 months
Description: AEs with onset in Part 1 that are ongoing in Part 2 were not included in the count of AEs in Part 2. Safety Population and OLE Safety Population were assessed. As pre-specified in study design, participants in Part 2 received individualized optimized treatment (0.2 mg/kg/day to 0.8 mg/kg/day) based on Investigator discretion. Hence overall data for Part 2 is reported.
Groups:
- Part 1: Cohort A- Placebo: Participants received matching placebo as an oral solution, twice a day (bid) over 2 weeks of Titration Period and an additional 12 weeks of Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days.
- Part 1: Cohort A- ZX008 0.2 mg/kg/Day: Participants received ZX008 0.2 milligram per kilogram per day (mg/kg/day) during the 2-week Titration. Following titration, participants received ZX008 0.2 mg/kg/day as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days.
- Part 1: Cohort A- ZX008 0.8 mg/kg/Day: Participants were titrated to their blinded randomized dose of ZX008 over the 2-week Titration from 0.2 mg/kg/day to ZX008 0.8 mg/kg/day (or a maximum dose of 30 mg/day or 20 mg/day for participants taking concomitant stiripentol [STP]). Following titration, participants continued to receive the randomized dose of ZX008 as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days.
- Part 1: Cohort B- Placebo: Participants received matching placebo as an oral solution, bid over 2 weeks of Titration Period and an additional 12 weeks of Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days.
- Part 1: Cohort B- ZX008 0.2 mg/kg/Day: Participants received ZX008 0.2 mg/kg/day during the 2-week Titration. Following titration, participants received ZX008 0.2 mg/kg/day as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days.
- Part 1: Cohort B- ZX008 0.8 mg/kg/Day: Participants were titrated to their blinded randomized dose of ZX008 over the 2-week Titration from 0.2 mg/kg/day to ZX008 0.8 mg/kg/day (or a maximum dose of 30 mg/day or 20 mg/day for participants taking concomitant STP). Following titration, participants continued to receive the randomized dose of ZX008 as an oral solution, bid for an additional 12 weeks during Maintenance Period. Participants who completed the Maintenance Period and did not continue in Part 2, and participants who discontinued from Part 1 early, were tapered off study medication over 8 days.
Arm/Group | Part 1: Cohort A- Placebo | Part 1: Cohort A- ZX008 0.2 mg/kg/Day | Part 1: Cohort A- ZX008 0.8 mg/kg/Day | Part 2: Cohort A- Overall | Part 1: Cohort B- Placebo | Part 1: Cohort B- ZX008 0.2 mg/kg/Day | Part 1: Cohort B- ZX008 0.8 mg/kg/Day | Part 2: Cohort B- Overall
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/89 | 1/87 | 1/247 | 0/11 | 0/11 | 0/11 | 0/32
Serious Adverse Events (participants affected / at risk) | 4/87 | 4/89 | 10/87 | 41/247 | 1/11 | 1/11 | 0/11 | 6/32
Other Adverse Events (participants affected / at risk) | 60/87 | 64/89 | 68/87 | 166/247 | 8/11 | 10/11 | 7/11 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort A- Placebo (N=87) | Part 1: Cohort A- ZX008 0.2 mg/kg/Day (N=89) | Part 1: Cohort A- ZX008 0.8 mg/kg/Day (N=87) | Part 2: Cohort A- Overall (N=247) | Part 1: Cohort B- Placebo (N=11) | Part 1: Cohort B- ZX008 0.2 mg/kg/Day (N=11) | Part 1: Cohort B- ZX008 0.8 mg/kg/Day (N=11) | Part 2: Cohort B- Overall (N=32)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden unexplained death in epilepsy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change in seizure presentation (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 8 (25) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stereotypy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoconus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication of device insertion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood prolactin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort A- Placebo (N=87) | Part 1: Cohort A- ZX008 0.2 mg/kg/Day (N=89) | Part 1: Cohort A- ZX008 0.8 mg/kg/Day (N=87) | Part 2: Cohort A- Overall (N=247) | Part 1: Cohort B- Placebo (N=11) | Part 1: Cohort B- ZX008 0.2 mg/kg/Day (N=11) | Part 1: Cohort B- ZX008 0.8 mg/kg/Day (N=11) | Part 2: Cohort B- Overall (N=32)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5) | 8 (10) | 18 (22) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 10 (10) | 10 (11) | 13 (15) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 5 (5) | 11 (16) | 9 (44) | 13 (17) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (5) | 4 (4) | 5 (5) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (11) | 8 (10) | 16 (18) | 33 (35) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 11 (13) | 11 (12) | 9 (10) | 25 (33) | 1 (1) | 0 (0) | 0 (0) | 7 (12)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 12 (14)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 8 (10) | 4 (5) | 7 (8) | 31 (43) | 2 (2) | 2 (2) | 0 (0) | 9 (18)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (10) | 6 (7) | 16 (20) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 5 (5) | 7 (10) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Blood prolactin increased (Investigations) | 1 (1) | 0 (0) | 3 (4) | 9 (10) | 0 (0) | 1 (1) | 0 (0) | 8 (14)
Echocardiogram abnormal (Investigations) | 6 (6) | 2 (2) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 2 (2) | 3 (3) | 7 (7) | 12 (12) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 13 (15) | 18 (18) | 32 (35) | 39 (42) | 2 (2) | 3 (4) | 3 (3) | 4 (4)
Change in seizure presentation (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 17 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 4 (4) | 5 (5) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 11 (13) | 5 (6) | 24 (28) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure cluster (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (5)
Somnolence (Nervous system disorders) | 10 (10) | 10 (11) | 15 (16) | 24 (26) | 1 (1) | 4 (5) | 3 (3) | 11 (16)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 3 (3) | 1 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Irritability (Psychiatric disorders) | 5 (5) | 9 (9) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 4 (4) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (5):
  • Study Protocol (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03355209/Prot_000.pdf
  • Statistical Analysis Plan: Part 2 Cohort B-SAP (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03355209/SAP_004.pdf
  • Statistical Analysis Plan: Part 2 Cohort A-SAP (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03355209/SAP_005.pdf
  • Statistical Analysis Plan: Part 1 Cohort B-SAP (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03355209/SAP_006.pdf
  • Statistical Analysis Plan: Part 1 Cohort A-SAP (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03355209/SAP_007.pdf